CLINICAL TRIAL: NCT04001270
Title: Core Cerebrospinal Fluid Biomarker Profile in Leucine Rich Glioma Inactivated 1 (LGI1) Antibody Associated Encephalitis
Brief Title: Core Cerebrospinal Fluid Biomarker Profile in Anti-Leucine Rich Glioma Inactivated 1 (Anti-LGI1) Encephalitis
Acronym: LGI1biom
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: LGI1biom
Record Dates: First submitted 2019-05-16; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Encephalitis; LGI1 Antibody Associated Encephalitis
Keywords: LGI1 encephalitis; Biomarkers; Cerebrospinal Fluid (CSF); Neurology
MeSH Terms: conditions — Encephalitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients anti leucine rich glioma inactivated-1 encephalitis: Biomarkers from patients with anti-leucine rich glioma inactivated 1 encephalitis (anti LGI1-E) will be studied. This is a non-interventional study involving biological samples (CSF biomarkers) already stored in biobank repositories. All stored samples were collected as part of the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population.

SUMMARY:
Limbic encephalitis associated with anti leucine-rich glioma inactivated-1 LGI1 antibody (anti-LGI1) usually presents with seizures and progressive disturbance of memory and behavior. But anti-LGI1 associated encephalitis (LGI1-E) could present with a variety of features including an elective cognitive form of the disease, which mimicks a neurodegenerative condition such as Creutzfeld Jakob disease or rapidly progressive Alzheimer disease. In these patients, the appropriate diagnosis could be challenging.

The primary aim of this study is to describe cerebrospinal fluid biomarkers in a cohort of LGI1-E patients as results of these markers are currently not described in LGI1-E. Moreover, patients with LGI1-E often present seizures. At this point, the impact on cerebrospinal fluid biomarkers has not been described in this condition. The secondary aims of this study are to compare cerebrospinal fluid (CSF) biomarkers in LGI1-E patients to these in other neurodegenerative conditions ( e.g. creutzfeld Jakob disease, Alzheimer disease), which are considered as a possible differential diagnosis in these patients. The last aim of this study is to look for correlations between cerebrospinal fluid biomarkers in LGI1-E and clinical data in these patients, especially seizure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of well characterized leucine rich glioma inactivated 1 (LGI1) antibody in serum or cerebrospinal fluid (CSF);
* LGI1 antibody associated encephalitis diagnosis according to the international guidelines;
* At least one core CSF biomarkers sample (T-tau, P-tau, AB-1-42) available after disease onset;
* Age at least 18 years old.

Exclusion Criteria:

* Absence of clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with leucine rich glioma inactivated 1 (LGI1) antibody associated encephalitis whose sample was sent for analysis at Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, for LGI1 antibody study and then stored at the biobank Neurobiotec
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-08-15 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Biomarker levels of leucine rich glioma inactivated 1 associated encephalitis | 3 months
  Core CSF biomarkers (T-tau, P-tau, Amyloid β Protein Fragment 1-42 (AB1-42), AB1-40, Neurofilament light chain, in ng/L) will be assessed in LGI1-E patients and will be compared to the profile of patients presenting with common and rapid Alzheimer's disease and with Creutzfeldt Jacob disease (CJD).
  For each biomarker, statistical comparisions will be made by Kruskal Wallis test then if needed with Wilcoxon Mann Whitney test.
Biomarker levels of anti leucine rich glioma inactivated 1 associated encephalitis | 3 months
  Neopterin Cerebrospinal Fluid (CSF) levels (nanomole/Liter, nmol/L) will be assessed in anti Leucine-rich Glioma inactivated-1 Encephalitis (LGI1-E) patients.
Biomarker levels of anti leucine rich glioma inactivated 1 associated encephalitis | 3 months
  Prion protein Cerebrospinal Fluid (CSF) levels (ug/L) will be assessed in LGI1-E patients

SECONDARY OUTCOMES:
Comparison of biomarker profile (T-tau, P-tau, Amyloid β Protein Fragment 1-42 (AB1-42), AB1-40, Neurofilament light chain, in nanograms/Liter (ng/L) | two weeks
  Statistical comparisons of CSF biomarker levels of patients presenting with anti leucine rich glioma inactivated 1 associated encephalitis with or without epileptic seizures. Mean comparisons will be made for each biomarker, with the Wilcoxon Mann Whitney test.
Comparison of biomarker profile in anti leucine rich glioma inactivated 1 associated encephalitis (LGI1-E) with versus without faciobrachial dystonic seizures. | two weeks
  Statistical comparisons of CSF biomarker levels of patients presenting with anti leucine rich glioma inactivated 1 associated encephalitis (LGI1-E) with or without faciobrachial dystonic seizures. Mean comparisons will be made for each biomarker, with the Wilcoxon Mann Whitney test.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie DESESTRET, Principal Investigator — Hospices Civils de Lyon